CLINICAL TRIAL: NCT02716350
Title: A Double Blind, Placebo Controlled, Randomised, Single Centred, Parallel Study to Determine the Potential of B-GOS, to Beneficially Influence the Wellbeing and Ageing in Healthy 52-65 Years Old Individuals
Brief Title: Effect of B-GOS on the Wellbeing and Ageing in Healthy 52-65 Years Old Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clasado Limited (Industry)
Collaborators: General Hospital, States of Jersey (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AGE2016
Record Dates: First submitted 2016-03-15; First posted 2016-03-23 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Healthy
MeSH Terms: interventions — maltodextrin; Starch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B-GOS (Experimental): powder, 3.5g/day
  Interventions: Dietary Supplement: B-GOS
- Maltodextrin (Placebo Comparator): powder, 3.5g/day
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: B-GOS — comparison versus placebo
  Other Names: Bimuno
  Arms: B-GOS
Dietary Supplement: Maltodextrin — placebo
  Other Names: corn starch
  Arms: Maltodextrin

SUMMARY:
To investigate the potential of B-GOS to beneficially influence the wellbeing and ageing in healthy adults (52-65 years old). The study will consist of a 4 month randomised double blind parallel treatment period with either B-GOS of Placebo, and 1 month follow up period without treatments.

DETAILED DESCRIPTION:
With age, several important alterations occur within the gastrointestinal (GI) tract, that are responsible for altered microbial environment (e.g. reduced diversity and number of beneficial bifidobacteria and higher populations of enterobacteria and clostridia).

Research over the past two decades has provided evidence that administration of probiotics (live microorganisms which, when administered in adequate amounts, confer a health benefit on the host) could be used to optimise gut microbiota and prevent and treat a range of diseases, as well as enhance immune function. Somewhat less documented and more recent concept is the use of prebiotics (nondigestible food ingredients that beneficially affect the host by selectively stimulating the growth and/or activity of one, or a limited number of bacteria in the colon). Prebiotics are naturally available in breast milk and in certain vegetables but can also be synthetic oligosaccharides of which the best known and the most researched examples include fructooligosaccharides (FOS) and galactooligosaccharides (GOS). B-GOS is a low molecular weight GOS mixture, shown to increase the number of probiotic bacteria, especially bifidobacteria, in younger and older adults, irritable-bowel sufferers and overweight adults. B-GOS also significantly decreases the colonisation and pathology of salmonellosis and incidence and duration of traveller's diarrhoea.

Our aim is to investigate the potential of B-GOS to beneficially influence the wellbeing and ageing in healthy adults (52-65 years old). The assessment would consist of various questionnaires covering quality of life, bowel function, mood and sleep and blood markers of inflammation and ageing.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 52 and 65 years of age
* In good general health, defined as no comorbidities requiring regular medical follow up
* Ability to communicate well with the investigator and to comply with the requirements of the entire study
* The volunteer has given written informed consent to participate and is willing to participate in the entire study

Exclusion Criteria:

* History or evidence of organic disease of the gastrointestinal tract; such as tumour, irritable bowel syndrome, etc., within the previous 5 years
* Consumed probiotic or prebiotic preparations on a regular basis (at least 3 times per week) in the last 2 weeks and during the trial period
* Former participation in another study involving prebiotic or probiotic preparations or investigational drugs within the previous 6 months, or intention to use such drugs during the course of the study
* Undergone surgical resection of any part of the bowel
* History of malignancy within the previous 5 years (with exception of well-treated basal cell carcinoma or in situ cervical carcinoma).
* Currently prescribed immunosuppressive drugs
* Intention to use regularly other medication which affects gastrointestinal motility and/or perception
* Current or recent history (within 12 months) of significant drug or alcohol abuse or dependence

Ages: 52 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-03; Primary Completion 2018-03 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
questionnaire as a measure of life quality | change from baseline answers to 4 (end of treatment) and 5 months (end of follow up)
  health related questions
C- reactive protein (CRP) | change from baseline CRP to 2, 4 (end of treatment) and 5 months (end of follow up)
  CRP will be measured by Ortho Diagnostics analyser from blood

SECONDARY OUTCOMES:
α1-antitrypsin | change from baseline α1-antitrypsin to 2, 4 (end of treatment) and 5 months (end of follow up)
  α1-antitrypsin will be measured by Ortho Diagnostics analyser from blood
blood pressure | measured monthly for 5 months
questionnaire as a measure of bowel function | measured monthly for 5 months
  diary that includes 5-consecutive days of questions related to stool frequency and consistency
questionnaire as a measure of mood | measured monthly for 5 months
  questions related to mood and sleep patterns
lipids | change from baseline lipids to 2, 4 (end of treatment) and 5 months (end of follow up)
  lipids will be measured by Ortho Diagnostics analyser from blood
glucose | change from baseline glucose to 2, 4 (end of treatment) and 5 months (end of follow up)
  glucose will be measured by Ortho Diagnostics analyser from blood
telomere shortening | change from baseline length of telomeres to end of the treatment period (4 months)
  telomeres will be measured from peripheral blood mononuclear cells

CONTACTS AND LOCATIONS:
Overall Officials: Jelena Vulevic, phd, Study Chair — Clasado Research Services
Locations (1):
- General Hospital Jersey, Saint Helier, Jersey, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
once the study is competed, codes will be unblinded and participants can receive their individual data upon written request - this is all listed in their information leaflets